CLINICAL TRIAL: NCT05950932
Title: Effects of Melissa Extract in Phytosome on Sleep Quality and Duration
Brief Title: Effects of Melissa Extract on Sleep Characteristics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Urbino "Carlo Bo" (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Davide Sisti, PhD, University of Urbino "Carlo Bo"
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UniUrb_Melissa_2023
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Sleep Disorder; Anxiety; Quality of Life
Keywords: sleep quality; quality of life; plant extract; melissa officinalis
MeSH Terms: conditions — Sleep Wake Disorders; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The treatment order (Melissa phytosome or placebo) will be randomly assigned using a binary random sequence generated through appropriate programming on an electronic spreadsheet. The order of phytosome/placebo administration will be achieved through block randomization (block size = 4), with participant stratification based on gender.
Who Masked: Participant, Investigator
Masking Description: The participants and the evaluators enrolling the participants will be blinded to the treatment conditions. The verum and placebo products will be packaged in indistinguishable separate containers, labeled with alphanumeric codes, and placed inside a dedicated kit. The alphanumeric keys related to the classification of products as treated/placebo will only be made available to the researchers after the data processing has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-Placebo (Experimental): This arm will assume firstly the supplement product (Melissa phytosome) and later the placebo.
  Interventions: Dietary Supplement: Melissa phytosome; Other: Placebo
- Placebo-Treatment (Experimental): This arm will assume firstly the placebo and later the supplement product (Melissa phytosome).
  Interventions: Dietary Supplement: Melissa phytosome; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melissa phytosome — Melissa phytosome® is composed of dry extract of Berberis aristata root (550mg/cpr), complexed with phospholipids (soy lecithin), Pisum sativa proteins, and proanthocyanidin oligomers from Vitis vinifera. 2 tablets of 200 mg Melissa phytosome will be provided to participants, to be taken 30 minutes before bedtime for 14 days.
Other: Placebo — 2 tablets with an equivalent form, color, flavor, and coating as the experimental product, to take 30 minutes before bedtime.

SUMMARY:
The plant Melissa officinalis L. is commonly used to treat disorders related to anxiety and sleep quality. It contains several phytochemicals that give it antioxidant, anti-inflammatory, antispasmodic, antimicrobial, and neuroprotective properties. A study on subjects with mild to moderate anxiety and sleep disorders showed that an extract of Melissa officinalis reduced anxiety manifestations by 18%, improved symptoms associated with anxiety by 15%, and reduced insomnia by 42%. However, that study did not have a control group, so a randomized trial with a control group is needed. The objective of the study will be to evaluate the beneficial effects of a phytosome-formulated Melissa officinalis extract on sleep duration and different stages of sleep, which will be monitored using a wrist device. She will be provided with a wrist device that will be used for sleep monitoring. The trial will last for 45 days, in which she will be asked to take the phytosome-formulated Melissa supplement for two 14-day periods (2 tablets, 30 minutes before bedtime). There will be a 7-day break in the intake period between the two periods. At the beginning, middle, and end of the trial, you will be asked to answer some questionnaires.

DETAILED DESCRIPTION:
Melissa officinalis L. is a plant belonging to the Lamiaceae family known for its beneficial properties. This plant has been used since ancient times to treat various disorders, especially those related to anxiety and sleep quality. M. officinalis contains several phytochemicals, such as phenolic acids, flavonoids, terpenoids, and many others, which form the basis of its pharmacological activities. The plant exhibits antioxidant, anti-inflammatory, antispasmodic, antimicrobial, and neuroprotective effects. Widely used since ancient times, M. officinalis has also been studied clinically, demonstrating interesting beneficial properties in the treatment of various conditions, including anxiety, sleep disorders, palpitations, hypertension, and depression. Nutraceuticals could be an alternative option to prescription drugs for alleviating symptoms associated with mild anxiety and insomnia. M. officinalis has been shown to be a stress-reducing and anxiolytic agent; in a study [Cases et al., 2011] conducted on subjects with mild to moderate anxiety and sleep disorders, M. officinalis extract reduced anxiety manifestations by 18%, improved anxiety-related symptoms by 15%, and reduced insomnia by 42%. Among the subjects who benefited from M. officinalis extract, 70% experienced a significant reduction in anxiety and 85% in insomnia. However, a limitation of the study was the absence of a control group, thus requiring a randomized controlled study with a placebo group. In light of the above, the aim of the current study is to further investigate the beneficial effects of a formulated M. officinalis extract in phytosome form (Phytosome®). The phytosome technology utilizes phospholipids derived from sunflowers as an element capable of modulating the absorption kinetics of plant-derived molecules, with the intention of optimizing the product's efficacy with the lowest effective dosage. The phytosome technology represents a potentially useful approach in optimizing the administration of M. officinalis extract, applicable to the described literature-based applications. Phytosome® is composed of a dry extract of Berberis aristata root (550mg/cpr), complexed with phospholipids (soy lecithin), Pisum sativa proteins, and proanthocyanidin oligomers from Vitis vinifera. The Melissa Phytosome-based product used has been registered with the Italian Ministry of Health. The specific application of interest is the induction and enhancement of physiological sleep dynamics.

The primary objective is to assess the duration of sleep using specific wearable devices, quantifying total sleep duration as well as the duration of deep sleep, light sleep, and REM (rapid eye movement) sleep. Sleep monitoring will be performed using the Garmin VenuSQ wrist device, a wearable smartwatch to be worn on the left wrist during the day and throughout the sleep monitoring period. The data will be recorded by the Garmin Connect application (Garmin Ltd), which monitors sleep duration in different phases and allows for data extraction. The devices will be provided to the participants by the recruiting center for the duration of the entire study (6 weeks; 5 weeks of study plus 1 week of training). The device enables the extraction of sleep phase durations for each subject at the end of the study [Burgett et al., 2019].

The secondary objectives are:

1. Monitoring subjective perceptions of sleep quality using the Insomnia Severity Index (ISI), a validated psychometric instrument for assessing the severity of nocturnal components of insomnia. It is often used as a measure of treatment response in clinical research.
2. Assessing perceived anxiety levels using the State-Trait Anxiety Inventory (STAI), a validated psychometric questionnaire consisting of 40 items on a Likert scale. The STAI measures two types of anxiety: state anxiety and trait anxiety.
3. Evaluating the improvement in quality of life using the Clinical Global Impression-Improvement scale (CGI-I), which is used to measure the improvement in quality of life associated with sleep disorder improvement. The CGI-I assesses the overall improvement of a subject's symptoms compared to baseline, with scores ranging from 1 (''very much improved'') to 7 (''very much worse'').
4. Monitoring any adverse effects using the DOTES scale. The DOTES considers 33 symptoms collected into six clusters (behavior and/or psychiatric symptoms, laboratory findings, neurological symptoms, neuro-vegetative symptoms, cardiovascular symptoms, and other symptoms), evaluated using Likert scales.

Allocation of Sleep Monitoring Devices The devices will be configured to create a remote-accessible account for each participant, allowing researchers to record sleep-related data. The devices will be collected at the end of the monitoring period and, after an appropriate reset and reconfiguration process, will be assigned to new subjects for monitoring.

Allocation of Nutraceutical Preparations

The verum and placebo products will be packaged in indistinguishable separate containers, labeled with alphanumeric codes, and placed inside a dedicated kit. Each kit should contain 14 doses consisting of either 2 tablets of 200 mg Melissa phytosome or 2 tablets with an equivalent form, color, flavor, and coating. The evaluated subjects will be instructed to take the 2 tablets 30 minutes before bedtime according to the following schedule:

* 14 days of kit 1 use
* 7-day washout period
* 14 days of kit 2 use

The assessment questionnaires will be administered via a computerized platform with the following timelines:

* T0
* T15
* T36

The alphanumeric keys related to the classification of products as treated/placebo will only be made available to the researchers after the data processing has been completed."

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Diagnosis of insomnia or sleep disturbances anxiety-related, since at least 30 days.

Exclusion Criteria:

* Breastfeeding
* Intention to become pregnant during the course of the study
* Consumption of anxiolytics, antidepressants, hypnotics, or sedatives within 10 days prior to the start of the study
* Diabetes
* Asthma
* Hypo- and hyperthyroidism
* Diagnosis of psychiatric and neurological disorders
* Treatment with psychotropic medications
* Treatment with antihistamines
* Alcoholism
* Smoking
* Current or past use of narcotics
* Use of melatonin
* Use of herbal remedies for sleep disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Sleep duration (hours and minutes) | From Day 0 to Day 36
  The sleep duration will be assessed as primary outcome, considering the total sleep time and the time spent in different sleeping phases.

SECONDARY OUTCOMES:
Perceived sleep quality (score) | Day 0, Day 15, Day 36.
  Perceived sleep quality usign the Insomnia Severity Index.
Perceived Anxiety (score) | Day 0, Day 15, Day 36
  Perceived anxiety levels using the State-Trait Anxiety Inventory (STAI).
Quality of life (score) | Day 0, Day 15, Day 36
  Perceived quality of life using the Clinical Global Impression-Improvement (CGI-I).
Adverse symptoms (number and severity) | From Day 0 to Day 36.
  Monitoring of possible adverse symptoms during the study, using the DOTES scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Urbino Carlo Bo, Urbino, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participants' data will be anonymized before sharing the collected data with other researchers in the research group.

REFERENCES:
- [Background] Cases J, Ibarra A, Feuillere N, Roller M, Sukkar SG. Pilot trial of Melissa officinalis L. leaf extract in the treatment of volunteers suffering from mild-to-moderate anxiety disorders and sleep disturbances. Med J Nutrition Metab. 2011 Dec;4(3):211-218. doi: 10.1007/s12349-010-0045-4. Epub 2010 Dec 17. PMID 22207903